CLINICAL TRIAL: NCT00772148
Title: A Phase 2, Open-Label, Multi-Center, Randomized Trial to Demonstrate the Pharmacokinetics of LCP-Tacro™ Tablets Once Daily and Prograf® Capsules Twice Daily in Adult De Novo Liver Transplant Patients
Brief Title: Pharmacokinetics of LCP-Tacro™ Once Daily and Prograf® Twice A Day in Adult De Novo Liver Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other); Aptuit (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCP-Tacro 2018
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Liver Failure
Keywords: Liver; Hepatic; Transplantation; Immunosuppression; Tacrolimus; Prograf
MeSH Terms: conditions — Liver Failure | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCP-Tacro (Experimental): LCP - Tacro™ tablets, once daily (LifeCycle Pharma A/S, Hørsholm DK)
  Interventions: Drug: LCP -Tacro
- Prograf (tacrolimus) (Active Comparator): Prograf® capsules, twice daily (Astellas Pharma US, Deerfield IL)
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: LCP -Tacro — LCP-Tacro tablets will be administered orally once daily in the morning starting at 0.07 - 0.11 mg/kg. The starting dose for African-American patients will be 0.09 - 0.13 mg/kg. Subsequent doses of each study drug will be adjusted to maintain target whole blood tacrolimus trough levels of 5 - 20 ng/mL.
  Other Names:Tacrolimus modified-release LCP-Tacro™ tablets (0.5 mg, 1 mg, 2 mg, 5 mg)
  Other Names: tacrolimus
  Arms: LCP-Tacro
Drug: Prograf — Oral Prograf capsules will be administered starting at 0.10 - 0.15 mg/kg per day in two equally divided morning and evening doses. Subsequent doses of each study drug will be adjusted to maintain target whole blood tacrolimus trough levels of 5 - 20 ng/mL.
  Other name: tacrolimus Prograf® capsules (0.5 mg, 1 mg, 5 mg)
  Other Names: tacrolimus
  Arms: Prograf (tacrolimus)

SUMMARY:
The purpose of this study is to demonstrate the pharmacokinetics (PK, measuring the amount of medication in blood samples) and safety of a new medicine, LCP-Tacro™ tablets, and Prograf® capsules, a drug commonly taken by transplant recipients to prevent the body from rejecting a transplanted kidney and liver. LCP-Tacro is a tablet containing the same active ingredient (tacrolimus) that is in Prograf capsules, but the tablet has been designed to release tacrolimus over an extended period so that it only has to be taken once daily. LCP-Tacro is an investigational drug.

This study will evaluate the levels of tacrolimus in the blood in the first two weeks after a liver transplant in patients randomly assigned (by chance, like flipping a coin) to take either LCP-Tacro™ tablets (tacrolimus) once daily or Prograf® capsules twice daily. In addition, patients will remain on study drug for 360 days in order to evaluate the relative safety of LCP-Tacro™ tablets compared to Prograf over a longer period of time.

DETAILED DESCRIPTION:
This was a randomized, parallel-group, open-label, multicenter study in adult de novo liver transplant patients to demonstrate the pharmacokinetics and safety of once-daily treatment of LCP-Tacro tablets and twice-daily Prograf capsules in the first 2 weeks after live transplantation. The study also compared the efficacy and safety of LCP-Tacro and Prograf over an additional 50 weeks after liver transplantation. Eligible patients were randomized (1:1 ratio) within 72 hours after transplantation (graft reperfusion) to receive either: 1) LCP-Tacr tablets orally once daily (QD) in the morning, with an interval of 24 +/- 1 hours between dosed, starting at 0.07 to 0.11 mg/kg (the starting daily dose for African-American patients was 0.09 to 0.13 mg/kg), or 2) Prograf capsules in 2 equally divided morning and evening doses, starting at 0.10 to 0.15 mg. Subsequent doses of study medications were to be adjusted by the investigator according to local practice to maintain a target whole blood tacrolimus trough level of 5 to 20 ng/mL thought Day 14. Twenty-four-hour pharmacokinetic assessments were performed on Days 1, 7 and 14; additionally whole blood tacrolimus trough levels for statistical analysis were measured on Days 2, 3, 4, 7, 10, 12, 12, 42, 90, 120, 180, 270, and 360. Physicians could also perform tacrolimus trough levels at other times at their discretion. On Day 360, the patients were placed on maintenance immunosuppressive regimen determined by their treating physician. Following completion of the third and final pharmacokinetic assessment on Day 14, patients entered the maintenance phase (Days 15 to 360) of study and remained on their assigned study medication until Day 360. Visits for safety assessments and tacrolimus trough levels during the maintenance phase were on Days 42, 90, 120, 180, 270 and 360.

Immunosuppressive therapy after the conclusion of the study was to be administered at the discretion of the patient's population.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women at least 18 years of age who are recipients of a liver transplant from a deceased donor with a Model for End-Stage Liver Disease (MELD) score at the time of transplantation of ≤ 30 who are able to give informed consent for participation

Exclusion Criteria:

* Recipient of any transplanted organ other than a liver
* Recipients of a liver from a non-heart beating donor
* Recipients of a liver from an ABO incompatible donor
* Recipients of a bone marrow or stem cell transplant
* Patients with a white blood cell count ≤ 2.8 x 109/L unless the absolute neutrophil count (ANC) is > 1.0 x 109/L
* Patients who fail a drugs of abuse screen in the pre-transplant evaluation
* Patients unable to swallow study medication
* Patients incapable of understanding the purposes and risks of the study, who cannot give written informed consent, or who are unwilling to comply with the study protocol
* Pregnant or nursing women (women of childbearing potential must have a negative serum pregnancy test within seven days prior to receiving study medication)
* Patients with reproductive potential who are unwilling/unable to use a double barrier method of contraception throughout the duration of the study
* Patients who were treated with any other investigational agent in the 30 days prior to enrollment
* Patients seropositive for human immunodeficiency virus (HIV)
* Patients with a current malignancy or a history of malignancy (within the past 5 years), except basal or non-metastatic squamous cell carcinoma of the skin that has been treated successfully, or hepatocellular carcinoma (HCC) that meet the Milan Criteria for liver transplantation
* Patients with uncontrolled concomitant infection, a systemic infection requiring treatment, or any other unstable medical condition that could interfere with the study objectives
* Patients with severe diarrhea, vomiting, active peptic ulcer or gastrointestinal disorder that may affect the absorption of tacrolimus
* Patients with a known hypersensitivity to tacrolimus
* Patients with any form of current substance abuse, psychiatric disorder or a condition that, in the opinion of the Investigator, may invalidate communication with the Investigator

Randomization to one of two treatment groups will be done post transplantation provided that the patient fulfills the following additional criteria:

* Patient is able to receive their first dose of randomized study drug orally within 72 hours after the transplant surgery (graft reperfusion)
* Patient was NOT given intravenous tacrolimus prior to their first oral dose of study medication
* Recipient of a liver with a cold ischemia time of ≤ 10 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angel Alsina, M.D., Principal Investigator — Tampa General Hospital, LifeLink Healthcare Institute
Locations (1):
- LifeLink Healthcare Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] DuBay DA, Teperman L, Ueda K, Silverman A, Chapman W, Alsina AE, Tyler C, Stevens DR. Pharmacokinetics of Once-Daily Extended-Release Tacrolimus Tablets Versus Twice-Daily Capsules in De Novo Liver Transplant. Clin Pharmacol Drug Dev. 2019 Nov;8(8):995-1008. doi: 10.1002/cpdd.657. Epub 2019 Jan 22. PMID 30667591

RESULTS

PARTICIPANT FLOW:
Groups:
- LCP-Tacro: LCP - Tacro™ tablets, once daily (LifeCycle Pharma A/S, Hørsholm DK)
  LCP -Tacro: LCP-Tacro tablets will be administered orally once daily in the morning starting at 0.07 - 0.11 mg/kg. The starting dose for African-American patients will be 0.09 - 0.13 mg/kg. Subsequent doses of each study drug will be adjusted to maintain target whole blood tacrolimus trough levels of 5 - 20 ng/mL.
  Other Names:Tacrolimus modified-release LCP-Tacro™ tablets (0.5 mg, 1 mg, 2 mg, 5 mg)
- Prograf (Tacrolimus): Prograf® capsules, twice daily (Astellas Pharma US, Deerfield IL)
  Prograf: Oral Prograf capsules will be administered starting at 0.10 - 0.15 mg/kg per day in two equally divided morning and evening doses. Subsequent doses of each study drug will be adjusted to maintain target whole blood tacrolimus trough levels of 5 - 20 ng/mL.
  Other name: tacrolimus Prograf® capsules (0.5 mg, 1 mg, 5 mg)
Period: Pharmacokinetic Phase (14 Days)
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Started | 29 | 29
Completed | 21 | 23
Not Completed | 8 | 6
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Administrative/other | 2 | 0
Period: Maintenance Phase (Week 52)
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Started | 21 | 23
Completed | 17 | 18
Not Completed | 4 | 5
Not completed — Death | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Administrative/other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCP-Tacro | Prograf (Tacrolimus) | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (7.27) | 54.6 (9.78) | 54.4 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 18
  Male | 24 | 16 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 24 | 27 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 2 | 4
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (Cmax and Cmin) of LCP-Tacro™ Compared to Prograf Early After Transplantations (Within the First 14 Days) in Adult de Novo Liver Transplant Recipients.
Description: The pharmacokinetic parameters (Cmax and Cmin) were evaluated during the first 14 days after liver transplant (on days 1, 7 and 14). The results for Day 14 is listed below as the primary outcome parameter for this study.
Time Frame: 14 days
Population: Arithmetic mean of the Pharmacokinetic parameters on Day 14 (mITT population)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Number analyzed (Participants) | 21 | 23
ng/mL
  Cmax | 21.30 (9.93) | 22.95 (14.57)
  Cmin | 7.41 (4.17) | 7.56 (2.64)

2. Secondary Outcome: Number of Participants Who Died Within the 360 Days.
Description: Number of patients who died was compared between the two groups during the study.
Time Frame: 360 days
Measure: Number; unit: participants
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Number analyzed (Participants) | 29 | 29
participants | 2 | 2

3. Primary Outcome: Pharmacokinetics (AUC0-24) of LCP-Tacro™ Compared to Prograf Early After Transplantations (Within the First 14 Days) in Adult de Novo Liver Transplant Recipients.
Description: The pharmacokinetic parameter (AUC, 0 to 24 hours post dose) was evaluated during the first 14 days after liver transplant (on days 1, 7 and 14). The results for Day 14 is listed below as the primary outcome parameter for this study.
Time Frame: 14 days
Population: Arithmetic mean of the Pharmacokinetic parameters on Day 14 (mITT population)
Measure: Mean (Standard Deviation); unit: ng/mL*hr
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Number analyzed (Participants) | 21 | 23
ng/mL*hr | 279.59 (139.86) | 241.22 (79.90)

4. Primary Outcome: Percentage of Patients in Each Treatment Group Achieving Sufficient Tacrolimus Whole Blood Trough Levels (5 to 20 ng/mL) During the First 14 Days Post-transplantation.
Description: Percentage of patients with trough levels within the therapeutic range of 5 to 20 ng/mL was assessed during the initial 14 days (on days 1, 7 and 14) after liver transplant and compared between the two treatment groups.
Time Frame: 1 day
Population: Percentage of patients achieving therapeutic tacrolimus trough levels on Day 1, Day 7 and Day 14.
Measure: Number; unit: percentage of patients
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Number analyzed (Participants) | 29 | 28
percentage of patients | 13.79 | 32.14

5. Primary Outcome: Percentage of Patients in Each Treatment Group Achieving Sufficient Tacrolimus Whole Blood Trough Levels (5 to 20 ng/mL) During the First 14 Days Post-transplantation.
Description: as for outcome 4
Time Frame: 7 days
Population: Percentage of patients achieving therapeutic tacrolimus trough levels on Day 1, Day 7 and Day 14.
Measure: Number; unit: percentage of patients
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Number analyzed (Participants) | 29 | 28
percentage of patients | 78.26 | 75

6. Primary Outcome: Percentage of Patients in Each Treatment Group Achieving Sufficient Tacrolimus Whole Blood Trough Levels (5 to 20 ng/mL) During the First 14 Days Post-transplantation.
Description: as for outcome 4
Time Frame: 14 days
Population: Percentage of patients achieving therapeutic tacrolimus trough levels on Day 1, Day 7 and Day 14.
Measure: Number; unit: percentage of patients
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Number analyzed (Participants) | 29 | 28
percentage of patients | 85.71 | 91.3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from date of first dose and until 30 days after last dose of study drug. For completing patients the collection time frame was 13 months.
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Serious Adverse Events (participants affected / at risk) | 17/29 | 10/29
Other Adverse Events (participants affected / at risk) | 29/29 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=29) | Prograf (Tacrolimus) (N=29)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardio-resiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Abdominla pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (4)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Aspargillosis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 2 (2) | 1 (1)
Incision site infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis Bacterial (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Woound infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Hepatitis C RNA positive (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyprglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bule duct cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=29) | Prograf (Tacrolimus) (N=29)
Anaemia (Blood and lymphatic system disorders) | 9 (13) | 9 (9)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Vission blurred (Eye disorders) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (11) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 10 (10) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 13 (17) | 11 (11)
Flatulence (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrooesophageal refluc syndrome (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (11) | 13 (13)
Vomiting (Gastrointestinal disorders) | 4 (7) | 5 (7)
Asthenia (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 8 (8) | 3 (3)
Generalised oedema (General disorders) | 2 (2) | 0 (0)
Oedema (General disorders) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 11 (14) | 10 (10)
Pain (General disorders) | 3 (4) | 2 (2)
Pyrexia (General disorders) | 5 (8) | 3 (4)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 2 (2)
Bile duct stenosis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 2 (5)
Jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0)
Liver transplant rejection (Immune system disorders) | 7 (8) | 5 (5)
Cystitis (Infections and infestations) | 0 (0) | 2 (2)
Hepatitis C (Infections and infestations) | 9 (9) | 8 (8)
Incision site infection (Infections and infestations) | 0 (0) | 2 (2)
Peritonitis bacterial (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (5)
Urinary tract infection (Infections and infestations) | 2 (3) | 4 (6)
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Complications of transplanted liver (Injury, poisoning and procedural complications) | 1 (1) | 2 (4)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Incision site pain (Injury, poisoning and procedural complications) | 1 (4) | 2 (2)
Post procedural bile leak (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (5) | 8 (9)
Skin laceration (Injury, poisoning and procedural complications) | 4 (7) | 4 (8)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 5 (7) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 2 (3)
Hepatic enzyme increased (Investigations) | 4 (4) | 4 (4)
Liver function test abnormal (Investigations) | 4 (6) | 5 (5)
Transaminases incrreased (Investigations) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Decreased apetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Fluid overload (Metabolism and nutrition disorders) | 7 (7) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (8) | 4 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (8) | 8 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (5) | 10 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 2 (3)
Headache (Nervous system disorders) | 10 (10) | 11 (12)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2) | 2 (2)
Tremor (Nervous system disorders) | 8 (8) | 10 (11)
Agitation (Psychiatric disorders) | 1 (1) | 2 (2)
Anxiety (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Confusional state (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Depression (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 1 (1)
Insomnia (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 6 (6)
Proteinurea (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (4) | 2 (2)
Renal failure acure (Renal and urinary disorders) | 2 (3) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 2 (2)
Scrotal oedema (Reproductive system and breast disorders) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Wheesing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (5) | 4 (4)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Post procedural drainage (Surgical and medical procedures) | 2 (7) | 1 (4)
Hypertension (Vascular disorders) | 3 (3) | 7 (7)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other